CLINICAL TRIAL: NCT04613349
Title: FArial NErf MRI in the Preoperative Assessment of PArotide Tumors
Acronym: NEFAPA
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 2020-A02019-30
Record Dates: First submitted 2020-07-07; First posted 2020-11-03 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Parotid Tumor
MeSH Terms: conditions — Parotid Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MRI — All patients included will benefit from the two methods of evaluating the anatomical relationships between the facial nerve and the parotid tumor:
  1. New medical imaging technique evaluated: high-resolution 3 Tesla parotid MRI with specific sequences and gadolinium injection;
  2. Gold standard: Intraoperative examination.

SUMMARY:
1. st visit: Inclusion, 3Tesla injected parotid MRI performed as part of routine care for characterization, to which two specific high resolution sequences will be added. Evaluation of the exact position of the parotid tumor relative to the trunk of the facial nerve and its first branches, classification into two categories: on contact (≤ 5 mm) or at a distance (> 5 mm).
2. nd visit: Surgical intervention of the parotid tumor. The surgeon will specify the same data as that collected by the radiologists after the MRI.
3. rd visit: Post-operative consultation in the week following the intervention. The surgeon will look for the occurrence of post-operative facial paralysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient candidate for first line surgery for a parotid tumor
* Parotid tumor located near the trunk of the facial nerve and or its first branches of division according to the clinical examination of the ENT surgeon and the imaging data
* Affiliate or beneficiary of a social security scheme
* Written consent to participate in the study

Exclusion Criteria:

* Personal history of parotid homolateral surgery
* Absolute or relative contraindication to MRI
* Known hypersensitivity to gadolinic contrast media
* Pre or post operative period of a liver transplant
* Patient benefiting from a legal protection measure
* Pregnant or lactating woman
* Patient who has already benefited from a preoperative MRI to characterize a complete, well conducted and interpretable parotid lesion

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient candidate for first line surgery for a parotid tumor
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2027-01-13 (Estimated); Study Completion 2027-05-13 (Estimated)

PRIMARY OUTCOMES:
measurements by the radiologist on the high resolution 3Tesla MRI with specific sequences. | day 0
  measurements by the radiologist on the high resolution 3Tesla MRI with specific sequences.
assessment by the surgeon during the excision surgery of the parotid lesion | day 0
  assessment by the surgeon during the excision surgery of the parotid lesion

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation A De Rothschild, Paris, PARIS, France

IPD SHARING:
Plan to Share IPD: No